CLINICAL TRIAL: NCT00947375
Title: The Effect of Lamictal TM Augmentation of Haloperidol Decanoate in the Treatment of Resistant Schizophrenia Predominantly by Verbal Resistant Hallucinosis: Randomized, Double-blind, Placebo-controlled, Study
Brief Title: Lamictal TM, Haloperidol Decanoate in Schizophrenia
Acronym: CMCOBaku
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: All of the mentioned aim and objectives were achieved before the February 2007
Sponsor: Central Mental Clinic for Outpatients of Baku City (Other)
Responsible Party: Chief Physician of Central Mental Clinic for Outpatients of Baku City, Chief Physician of Central Mental Clinic for Outpatients of Baku City
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Nadir
Record Dates: First submitted 2009-07-20; First posted 2009-07-28 (Estimated); Last update posted 2009-07-28 (Estimated); Status verified 2009-07

CONDITIONS: Schizophrenia
Keywords: schizophrenia; lamictal TM; haloperidol decanoate
MeSH Terms: conditions — Schizophrenia | interventions — haloperidol decanoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Starch (Experimental): In these study participants are randomly (by chance) assigned for two treatment arms of a clinical trial.
  Interventions: Drug: Lamictal TM; Drug: Haloperidol Decanoate
- Lifestyle councelling (No Intervention): May be required to comply with US Public Law 110-85, Section 801

INTERVENTIONS:
Drug: Lamictal TM — First group patients received either haloperidol deaconate 50 mg in weekly intramuscular and Lamictal TM 150-200 mg in day per so for 12 weeks.
  Arms: Starch
Drug: Haloperidol Decanoate — Second group patients were given haloperidol deaconate 50 mg in weekly intramuscular and placebo per os for 12 weeks.
  Arms: Starch

SUMMARY:
The purpose of this study is to determine the effect of lamotrigine augmentation of Haloperidol decanoate in the treatment of Resistant Schizophrenia predominantly by verbal resistant hallucinosis: A randomized, double-blind, placebo-controlled, study.

Nadir A.Aliyev & Zafar N.Aliyev

Central Mental Clinic for Outpatients of Baku city of Azerbaijan Republic

Abstract:

OBJECTIVE: The current paper reports on a double-blind, randomized study of the role of lamotrigine as an augmentation agent to haloperidol decanoate in the treatment of out patient's schizophrenia with verbal resistant hallucinosis.

DETAILED DESCRIPTION:
METHOD:A structured clinical interview, for DSM-IV Axis I Disorder, Patient Edition, was used to diagnose schizophrenia according to DSM-IV. Three hundred fifty patients were studied. The patients were then randomly divided into two groups on 175 subjects in each group. First group patients received either haloperidol deaconate 50 mg in weekly intramuscular and lamotrigine 150-200 mg in day per so for 12 weeks. Second group patients were given haloperidol deaconate 50 mg in weekly intramuscular and placebo per os for 12 weeks. Data for clinical assessments were collected at weeks 0, 6 and 12 weeks. The expressiveness of psychopathology was estimated on PANSS. Test response in both groups was defined as a reduction in the PANSS by using analysis of variance and chi-square tests.

ELIGIBILITY:
Exclusion Criteria:

* Display an acute systemic medical disorder or a medical disorder requiring frequent changes in medication;
* Display a history of seizures, cerebrovascular disease, structural brain damage, from trauma, focal neurological sings on examination, or evidence of any progressive neurological disorder, substance dependence (except tobacco).

Inclusion Criteria:

* age from 18-60;
* both gender;
* resistant scizophrenia patients;
* previous treatment history;
* verbal resistant hallucinosis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 335 (Actual)
Dates: Start 2005-01; Primary Completion 2006-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Data suggest that haloperidol decanoate with the combination of lamotrigine was more effective than placebo. | 2006

SECONDARY OUTCOMES:
lamotrigine augmentation of haloperidol decanoate improve treatment-resistant schizophrenia | 2007

CONTACTS AND LOCATIONS:
Overall Officials: Nadir A Aliyev, PHD, MD, Principal Investigator — Outpatient service
Locations (1):
- Central Mental Clinic for Outpatients of Baku City, Baku, Azerbaijan